CLINICAL TRIAL: NCT05772260
Title: Effect of Autonomic Dysfunction on Hemodynamic Instability During Per-oral Endoscopic Myotomy in Achalasia Patients: a Prospective Observational Study
Brief Title: Autonomic Dysfunction and Hemodynamic Instability During Per-oral Endoscopic Myotomy
Status: Recruiting | Type: Observational
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Dong Woo Han, Professor, Gangnam Severance Hospital
Other Study IDs: 3-2022-0491
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Achalasia
MeSH Terms: conditions — Esophageal Achalasia | interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with autonomic dysfunction: Achalasia patients who have autonomic dysfunction in the heart rate variability test (HRV test) performed preoperatively.
  Interventions: Procedure: Per-oral endoscopic myotomy
- Patients with normal autonomic function: Achalasia patients without autonomic dysfunction in the heart rate variability test (HRV test) performed preoperatively.
  Interventions: Procedure: Per-oral endoscopic myotomy

INTERVENTIONS:
Procedure: Per-oral endoscopic myotomy — Per-oral endoscopic myotomy will be performed under general anesthesia. Per-oral endoscopic myotomy will be performed according to the standard care.
  General anesthesia will be conducted according to the standard care in our institution, and standardized as follows.
  * Monitoring: ECG, SpO2, noninvasive blood pressure, invasive blood pressure monitoring via radial artery cannulation, advanced hemodynamic monitoring (including cardiac output, cardiac index) uisng EV1000 clinical platform (Edwards Lifesciences, USA), anesthetic depth monitoring by SedLine Sedation monitor (Masimo corporation).
  * Anesthetic induction: Target controlled infusion (TCI) of Remifentanil (target 3.0 ng/mL), propofol 2 mg/kg IV, rocuronium 0.8 mg/kg IV
  * Anesthetic maintence: sevoflurane 0.9 age corrected MAC and remifentanil TCI (target range 1.0-4.0 ng/mL)
  Other Names: general anesthesia

SUMMARY:
This prospective observational study aims to investigate the association between the autonomic dysfunction and hemodynamic instability during per-oral endoscopic myotomy under general anesthesia in achalasia patients. Per-oral endoscopic myotomy is known as the effective treatment for achalasia patients. During per-oral endoscopic myotomy, capnoperitoneum, capnomediastinum, and systemic CO2 accumulation can potentially impair hemodynamics. Moreover, it has been suggested that achalasia is associated with autonomic dysfunction. We hypothesized that patients with autonomic dysfunstion would esperience more hemodynamic instability during per-oral endoscopic myotomy compared with patients without autonomic dysfunction. In this prospective observational study, the autonomic function test will be performed before surgery, and advanced hemodynamic parameters will be recorded using EV1000 clinical platform (Edwards Lifesciences, USA) during surgery. The association between the autonomic dysfunction and hemodynamic instability during per-oral endoscopic myotomy will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are scheduled to undergo per-oral endoscopic myotomy in Gangnam Severance Hospital
2. Patients aged ≥ 19 years

Exclusion Criteria:

1. Patients who are hemodynamically unstable before surgery
2. Patients in whom preoperative heart rate variability (HRV) test cannot be conducted
3. Pregnant women of breastfeeding women
4. Patients unable to read the informed consent form

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who are scheduled to undergo per-oral endoscopic myotomy in Gangnam Severance Hospital will be eligible.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Wobble of Systolic Arterial Pressure (SAP) during surgery | During the intraoperative period, from the enterance to the operating room to the emergence of anesthesia
  Wobble of SAP will be calculated according to the following formula. Performance Error (PE (%)) = (measured SAP-reference SAP) × 100/reference SAP Median performance error (MDPE (%)) = median {PEi, i = 1, 2, 3…, N} Median absolute performance error (MDAPE (%)) = median {|PE| , i = 1, 2, 3…, N} (N, number of measured SAP) Wobble (%) = median{|MDPE - PEi|, i = 1, 2, 3…, N}(N, number of measured PE) reference SAP = 120 mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- GangnamSeverance Hospital, Seoul, South Korea

REFERENCES:
- [Background] Saugel B, Vokuhl C, Pinnschmidt HO, Rosch T, Petzoldt M, Loser B. Cardiovascular dynamics during peroral endoscopic myotomy for esophageal achalasia: a prospective observational study using non-invasive finger cuff-derived pulse wave analysis. J Clin Monit Comput. 2021 Aug;35(4):827-834. doi: 10.1007/s10877-020-00541-8. Epub 2020 Jun 5. PMID 32504156